CLINICAL TRIAL: NCT02401906
Title: MRI for the Etiological Diagnosis of Orbital Tumours
Brief Title: MRI and Orbital Tumours (MEDORT)
Acronym: MEDORT
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2015-8
Record Dates: First submitted 2015-03-17; First posted 2015-03-30 (Estimated); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Orbital Tumor; Orbital Pseudotumor
MeSH Terms: conditions — Orbital Neoplasms; Orbital Pseudotumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MRI

SUMMARY:
Orbital masses develop at the expense of the orbital structures lacrimal glands, oculomotor muscles, optic nerve, meningeal spaces, peripheral nerves, bone wall, orbital fat, lymphoid structures or vascular structures. These masses can be tumors, benign or malignant, or pseudotumor, mainly represented by specific or non-specific orbital inflammation.

Pathology is of considerable importance for the diagnosis and the treatment of those masses. However, biopsy or surgical resection of the orbital masses is sometimes difficult and dangerous outside expert centers.

The identification of a non-invasive technique for distinguishing tumors from pseudotumors, thus avoid in some cases a biopsy, would be a major contribution for the patients.

The MRI assessment performed routinely in a patient with an orbital mass includes morphological sequences T1, T2 fat suppression, T1 injected fat suppression, diffusion. This exploration requires, regardless of the performed research, a contrast agent injection (0.1 mg / kg weight of Gadobutrol®).

In this research protocol, during the injection of the contrast agent performed during the MRI assessment performed routinely, a DCE perfusion sequence, which consists of a repeated acquisition at short intervals of a volume gradient echo T1, will be added. This acquisition will be preceded by two short series for calibration. The post treatment will include parametric permeability cards (Ktrans) and plasmatic volume (Vp), evaluating one or more regions of interest in the tumor, normal lacrimal glands, jaw muscles and nasal mucosa being the reference. It will also be added a magnetic susceptibility EPI sequence type. All the qualitative parameters (T1, T2, T1 injected, distribution, low signal intensity in susceptibility) and quantitative (Ktrans, Vp, relative intensity enhancement, apparent diffusion coefficient) parameters will be collected.

The result of the pathological exam of the biopsy or of the surgical specimen, which is the gold-standard, will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years, with an orbital mass for which a biopsy or a resection is planned, coming for an MRI, before any surgical treatment

Exclusion Criteria:

* Absolute or relative contra-indication to MRI or to a contrast agent gadolinium injection (including pregnant or likely to be, breastfeeding women)
* Patient under guardianship
* Patient not willing to participate.
* Lack of affiliation to social security or medical state aid (AME) or universal health coverage (CMU)
* Motion artifact on the sequences, not corrected by the repeat sequences
* Metal artifact prohibiting the analysis of the region of interest
* Biopsy or resection not performed, particularly if the orbital mass is due to an infection
* MRI findings allowing a diagnosis without the need for pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged over 18 years, with an orbital mass for which a biopsy or a resection is planned, coming for an MRI, before any surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity based on the patterns of the intra voxel incoherent motion, the dynamic susceptibility contrast and enhancement, for distinguishing orbital tumors from orbital pseudotumor, the gold standard being the pathological exam. | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation ophtalmique Adolphe de Rothschild, Paris, France

REFERENCES:
- [Result] O'Shaughnessy E, Senicourt L, Mambour N, Savatovsky J, Duron L, Lecler A. Toward Precision Diagnosis: Machine Learning in Identifying Malignant Orbital Tumors With Multiparametric 3 T MRI. Invest Radiol. 2024 Oct 1;59(10):737-745. doi: 10.1097/RLI.0000000000001076. Epub 2024 Apr 11. PMID 38597586